CLINICAL TRIAL: NCT01724099
Title: A Double Blind, Randomized, Multicenter, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Euiiyin-tang on Obese Patients
Brief Title: Evaluating the Safety and Efficacy of Euiiyin-tang on Obesity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Korea Health Industry Development Institute (Other Government); Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Gyu Ko, Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP001
Record Dates: First submitted 2012-11-02; First posted 2012-11-09 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Obesity
Keywords: Obesity; Herbal product; Korean Medicine
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Euiiyin-tang (Experimental): powder type, 3 times per day before the meal, 12 weeks total
  Interventions: Drug: Euiiyin-tang
- Placebo (Placebo Comparator): powder type, 3 times per day before the meal, 12 weeks total
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Euiiyin-tang — Korean medicinal herbal drug
  Arms: Euiiyin-tang
Drug: Placebo — Placebo drug, same odor and formula as Euiiyin-tang
  Arms: Placebo

SUMMARY:
The hypothesis of this study is obese patient with Euiiyin-tang for 12 weeks will show a superior reduction compared to those taking the placebo.

DETAILED DESCRIPTION:
This study has two arms, Euiiyin-tang and placebo group. Inclusion of 80 patient each arm. They will be screened at first visit. At the baseline, that is the second visit, they will be evaluated each outcomes including weight, waist circumference, lipid profile (total cholesterol, triglyceride), CRP (C-reactive protein), visceral fat area and subcutaneous fat area using abdominal computed tomography (CT), questionnaires of QoL (Quality of Life) and eating attitudes, etc. The Euiiyin-tang will provide to the patients from the baseline, it contains 4 weeks of serving. After 4 weeks, the visit 3, the evaluation procedure will be repeated except lipid profile, CRP, abdominal CT. Another Euiiyin-tang of 4 weeks will be given to the patient. The visit 4, 4 weeks after the visit 3, the same procedure will be repeated. The visit 5, 12 weeks after from the baseline, the patient will be evaluated including weight, waist circumference, lipid profile, CRP, visceral fat area and subcutaneous fat area using abdominal computed tomography, questionnaires of QoL and eating attitudes, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-65 years old
2. Patients applying to one of the followings 2.1. BMI 30kg/m2 or over 2.2. BMI 27-29.9kg/m2 with hypertension in a proper treatment and blood pressure controlled (SBP ≤ 145mmHg, DBP ≤ 95mmHg) 2.3. BMI 27-29.9kg/m2 with non-insulin-dependent diabetes mellitus and fasting blood glucose < 7.8mmol/L(140mg/dL) 2.4. BMI 27-29.9kg/m2 with hyperlipidemia in a proper treatment 2.5. BMI 27-39.9kg/m2 and Total cholesterol 236mg/dL or over or Triglyceride 150mg/dL or over at screening
3. Agreed to low-calorie diet during the trial
4. Written informed consent of the trial

Exclusion Criteria:

1. Endocrine disease such as hypothyroidism, Cushing's syndrome, etc.
2. Heart disease (heart failure, angina pectoris, myocardial infarction)
3. Uncontrolled hypertension (SBP > 145 mmHg or DBP > 95 mmHg)
4. Malignant tumour or lung disease
5. Cholelithiasis
6. Severe renal disability (SCr > 2.0 mg/dL)
7. Severe liver disability (2.5 fold of normal high range value on Alanine Aminotransferase [ALT], Aspartate Aminotransferase [AST], alkaline phosphatase)
8. Non-insulin-dependent diabetes mellitus and fasting blood sugar 7.8mmol/L (140 mg/dL) or over
9. Narrow angle glaucoma
10. History or existence of neurological or psychological disease (schizophrenia, epilepsy, alcoholism, drug addiction, anorexia, bulimia, etc.)
11. History of stroke or temporary ischemic cardioplegia
12. History or existence of eating disorder such as anorexia nervosa or bulimia nervosa, etc.
13. Use of medication that could have effect on weight within last 3 months (appetite suppressant, laxative, oral steroid, thyroid hormone, amphetamine, cyproheptadine, phenothiazine or medication having effect on absorption, metabolism, excretion)
14. Use of β--blocker or diuretic as hypertension medication within last 3 months
15. Use of medication for central nervous system or central active weight reduction medication
16. Forbidden treatment (Insulin, hypoglycemic agent, antidepressant, antiserotonin agent, barbiturate, antipsychotic, medication concerns of abuse)
17. Difficult to measure anthropometric dimensions because of anatomical change such as resection
18. Surgical history for weight reduction; bariatric surgery, etc.
19. Unable to follow instructions of the trial as judged by investigator
20. Women who were pregnant, lactating, planning a pregnancy or women of childbearing age who do not agree to proper contraception (birth-control pill, hormone implant, IUD, spermicide, condom, abstinence, etc.) (Women of childbearing age indicate within 2 years of menopause who did not receive hysterectomy, bilateral tubal ligation, bilateral oophorectomy, etc.)
21. Use of other investigational product within last 1 month
22. Reduction over 10% of the previous weight within 6 months
23. Decided to stop smoking within last 3 months; however, keeping irregular smoking habit

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Weight reduction | between baseline and 12 weeks

SECONDARY OUTCOMES:
C-reactive protein (CRP) | baseline and 12 weeks
Blood pressure | baseline, 4 weeks, 8 weeks, and 12 weeks
Blood glucose | baseline and 12 weeks
Waist/hip ratio | 4 weeks, 8 weeks, and 12 weeks
Waist circumference | baseline, 4 weeks, 8 weeks, and 12 weeks
Korean Obesity-related Quality of Life scale | baseline and 12 weeks
Korean version of Eating Attitudes Test-26 | baseline and 12 weeks
Total cholesterol | baseline and 12 weeks
Triglyceride | baseline and 12 weeks
Visceral fat area | baseline and 12 weeks
  Using abdominal computed tomography
Subcutaneous fat area | baseline and 12 weeks
  Using abdominal computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-kyung SONG, KMD, Principal Investigator — Gachon University Medical Center
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

REFERENCES:
- [Derived] Cheon C, Song YK, Ko SG. Efficacy and safety of Euiiyin-tang in Korean women with obesity: A randomized, double-blind, placebo-controlled, multicenter trial. Complement Ther Med. 2020 Jun;51:102423. doi: 10.1016/j.ctim.2020.102423. Epub 2020 May 21. PMID 32507436
- [Derived] Cheon C, Jang S, Park JS, Ko Y, Kim DS, Lee BH, Song HJ, Song YK, Jang BH, Shin YC, Ko SG. Euiiyin-tang in the treatment of obesity: study protocol for a randomised controlled trial. Trials. 2017 Jun 21;18(1):289. doi: 10.1186/s13063-017-2039-8. PMID 28637494